CLINICAL TRIAL: NCT00963664
Title: Phase 2 Study of Interferon Alfa-2b and Lovastatin Combination Therapy for Patients With High-risk Resected or Unresectable Malignant Melanoma
Brief Title: Evaluation of Interferon-Lovastatin Therapy for Malignant Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Modifications will be necessary before full IRB approval will be secured.
Sponsor: NeoPlas Innovation (Other)
Responsible Party: Stephen B. Cantrell MD, Director of Research, NeoPlas Innovation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI-MM-009
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Melanoma; Malignant Melanoma
Keywords: melanoma; malignant melanoma; interferon; interferon alfa-2b; Intron-A; Intron A; Intron; lovastatin; mevinolin; Mevacor; statin; HRI
MeSH Terms: conditions — Melanoma | interventions — Lovastatin; Interferon alpha-2; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interferon and lovastatin treatment (Experimental): Patients receive outpatient treatment with lovastatin (oral) and interferon alfa-2b (subcutaneous injection) as per protocol parameters.
  Interventions: Drug: lovastatin; Drug: interferon alfa-2b

INTERVENTIONS:
Drug: lovastatin — lovastatin tablets, oral administration, daily dose 1.5 mg/kg, divided into three or four essentially equal doses with meals
  Other Names: Mevacor
Drug: interferon alfa-2b — interferon alfa-2b for subcutaneous injection, each injection 100,000 international units per kg body mass, three injections weekly
  Other Names: Intron-A

SUMMARY:
The purpose of this study is to determine whether an outpatient combination of lovastatin and low-to-moderate dose interferon is effective in the treatment of patients with malignant melanoma.

DETAILED DESCRIPTION:
Malignant melanoma, or simply melanoma, is a potentially fatal cancer which begins as a skin cancer and can spread very aggressively. The incidence of melanoma has been rising rapidly over the last decade and it is now becoming a serious health threat in young adults as well as older adults. Unfortunately, if melanoma escapes complete surgical removal, there are very few treatments which have been found very effective in controlling its growth and spread. If the cancer spreads to the lymph node system or beyond, the chances for long-term survival can be very poor.

This study proposes to test the effectiveness for melanoma treatment of a combination of two medicines which are in widespread use for other medical conditions. Interferon alfa-2b (also known simply as interferon or by a brand name Intron-A) is an exact replica of a protein produced by the human immune system. The human body makes this immune system regulator to help it kill cells in the body which are damaged or infected and thus need to be removed before they can cause further harm to the body. This medicine is often prescribed for infections like hepatitis, some types of cancer including melanoma, and immune system disorders. This study uses interferon in moderate doses, much less than typically used for melanoma treatment when it is used alone, and so the side effects of treatment may be milder. The other medicine being used in combination with it is lovastatin. This medicine is most often used to help patients reduce their cholesterol levels and therefore reduce the risk of heart attacks and strokes. Millions of people use this medicine because it has been found very safe and effective. Research has shown that it also has significant effects against the growth of cancer cells in laboratory cultures and in some animal models.

These two medicines have been used together to treat patients with cancer for several years in our medical practice, but until now they have not been formally tested in a clinical trial. This study will test how well the combination of these medicines can perform and test the hypothesis that they can achieve better survival and control of disease than currently available standard treatment. The incidence of side effects and other details will be monitored too.

This study is open to qualifying patients with stage 2, 3, or 4 melanoma. The results for patients in each group will be compared to other patients in the study with the same or similar stage of disease and with historical results of patients receiving the standard, already-approved treatments for similar stages of melanoma.

ELIGIBILITY:
Inclusion Criteria: (patients must meet all these criteria)

* Histologically confirmed diagnosis of malignant melanoma
* AJCC stage 2, 3, or 4 disease subject to the planned patient enrollment numbers for this trial
* Surgical resection to the extent possible
* ECOG performance status of 0, 1, or 2
* Expected survival of six months or greater
* ALT (SGPT) and AST (SGOT) not greater than 2.5x upper limit of normal range
* CT, PET or other valid imaging sufficient to demonstrate extent of disease performed less than three weeks prior to initiation or less than two weeks following initiation
* Female patients of childbearing potential must agree to practice contraception, abstinence, or other effective pregnancy avoidance measures while enrolled in this trial and for one month afterward

Exclusion Criteria: (patients meeting any of these criteria are ineligible)

* Current or anticipated pregnancy or breastfeeding
* History of or evidence suggestive of cerebral metastatic disease
* Impaired ability to absorb nutrition and/or medications normally via gastrointestinal tract
* Less than 18 years of age
* History or evidence of cirrhosis, chronic hepatitis, pancreatitis, or other significant hepatobiliary impairment
* History or evidence of HIV infection or other immune system impairment
* History of organ or tissue transplant requiring immunosuppressive therapy
* History of neutropenia other than that induced by chemotherapy
* Cytotoxic chemotherapy or radiation treatment within three weeks prior to initiation
* Presence of greater than six identifiable tumors counting all primary and metastatic lesions
* Presence of any single tumor mass greater than 6 cm in greatest dimension
* Presence of three or more tumor masses greater than 4 cm in greatest dimension
* Chronic steroid or immunosuppressive therapy
* Any other serious medical condition which, in the medical opinion of the investigator, limits life expectancy to two years or less or has significant potential for debilitation
* Any condition, psychiatric or otherwise, which may preclude valid informed consent or consistent compliance with study requirements in the medical opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2009-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 6 months, 1 yr, 2 yr, 3 yr, 4 yr, 5 yr
Time to progression of disease | 2 mos, 4 mos, 6 mos, 1 yr, 2 yr, 3 yr, 4 yr, 5 yr

SECONDARY OUTCOMES:
Appearance of new distant metastases | 2 mos, 4 mos, 6 mos, 1 yr, 2 yr, 3 yr, 4 yr, 5 yr
Toleration of medication side effects and quality of life | 4 mos, 1 yr, 2 yr, 3 yr, 4 yr, 5 yr

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B. Cantrell, MD, Principal Investigator — NeoPlas Innovation
Locations (1):
- NeoPlas Innovation, Nashville, Tennessee, United States